CLINICAL TRIAL: NCT05970068
Title: Implantation of Hydrophobic Tubes for Edema Fluid Drainage in Obstructive Lymphedema of Limbs - a Randomized Clinical Trial
Brief Title: Hydrophobic Tubes for the Treament of Lower and Upper Limb Lymphedema
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, MD, MPH, PHD, FEBVS, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300-23
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Lymphedema of Leg
Keywords: Lymphedema; quality of life; edema; lower limb
MeSH Terms: conditions — Lymphedema; Edema

STUDY DESIGN:
Intervention Model Description: Once eligible patients have been identified, they would be randomized into one of two groups - the intervention group or the control group.
  Randomization will help ensure that the two groups are comparable in terms of baseline characteristics, which can minimize the risk of bias in the study. The program used will be https://www.random.org/lists/.
  Group 1: Surgery + best medical treatment The intervention group would receive the novel treatment of implantation of hydrophobic tubes for edema fluid drainage, in addition to the best medical treatment available.
  Group 2: best medical treatment This control group would receive only the best medical treatment available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Surgery + best medical treatment (Experimental): The intervention group would receive the novel treatment of implantation of hydrophobic tubes for edema fluid drainage and the best medical treatment available.
  Interventions: Procedure: implantation of hydrophobic tubes for edema fluid drainage; Device: Best Medical Treatment
- Group 2: best medical treatment (Active Comparator): This control group would receive only the best medical treatment available.
  Interventions: Device: Best Medical Treatment

INTERVENTIONS:
Procedure: implantation of hydrophobic tubes for edema fluid drainage — 1 - A 2-cm-long incision is made at the border of the hypogastrium or lumbar region 10 cm above the inguinal crease; 2- A 1.5-cm-wide and 100-cm-long metal tube tunneling device is introduced under the skin and bluntly passed in the subcutaneous tissue toward the thigh and internal aspect of the calf; 3- Incisions 2 cm long are made in the groin and calf, through which the tunneling device was passed; 4-The hydrophobic tube is passed upward through the tunneling device, after which the tunneling device is removed; 5-The upper and lower ends of the hydrophobic tubes are fixed to the fascia with absorbable sutures.
  Arms: Group 1: Surgery + best medical treatment
Device: Best Medical Treatment — Compressive therapy, Phisioterapy, venous intervention

SUMMARY:
Lymphedema is a chronic condition causing fluid buildup in affected limbs. Traditional treatments often fall short, but subcutaneous implantation of hydrophobic silicone tubes shows promise, creating artificial drainage pathways. This approach proved effective in managing obstructive lymphedema in lower limbs. Further research is needed to validate its efficacy and explore long-term outcomes.

DETAILED DESCRIPTION:
Lymphedema is a chronic condition that affects the lymphatic system and accumulates protein-rich fluid in the interstitial spaces of the affected limb. The condition can occur after surgery, trauma, radiation therapy, or infection and can cause significant physical, functional, and psychosocial impairment. The chronic swelling and fibrosis of the affected limb can lead to difficulty with daily activities, decreased mobility, reduced quality of life, and increased susceptibility to infections (1).

Currently, the management of lymphedema involves both conservative and surgical approaches. Conservative treatment includes complex decongestive therapy, which combines manual lymphatic drainage, compression therapy, exercise, and skincare (reference here). While this approach can be effective, it requires long-term commitment and compliance from patients, which can be challenging (reference here). Surgical approaches, such as lymphaticovenular anastomosis or vascularized lymph node transfer, are reserved for patients with mild to severe or refractory lymphedema with moderate results (2).

Liposuction has been used as a treatment for lower limb lymphedema. The traditional treatment of lymphedema includes compression garments, exercise, and manual lymphatic drainage, but these methods are not very effective.

In advanced cases of lymphedema, where all main lymphatics vessels are obstructed, one possible solution may be to create artificial pathways for edema fluid to flow away from the obstructed regions. This can be achieved through the subcutaneous implantation of silicone tubes, a novel method for draining edema fluid in obstructive lymphedema of limbs (3).

In the lower limbs, the tubes are placed from the leg to the lumbar or hypogastric region, creating channels for fluid to flow away from the obstructed areas to the non-obstructed regions, where absorption can take place.

The subcutaneous implantation of hydrophobic tubes is a minimally invasive procedure that has shown promising results in the management of obstructive lymphedema of the lower limbs.

In a group of 20 patients with obstructive lymphedema of the lower limbs that developed after lymphadenectomy and irradiation of the pelvis because of uterine cancer, this procedure was found to be effective after unsuccessful conservative therapy. The patients underwent the implantation of hydrophobic silicone tubes, followed by external compression using intermittent pneumatic compression and elastic support of tissues (3).

Overall, the implantation of hydrophobic tubes presents a promising alternative for managing obstructive lymphedema of the lower limbs. It has the potential to improve the quality of life for those who suffer from this condition, especially in advanced cases where other treatment options have failed. Further research is necessary to validate the efficacy of this approach and its long-term outcomes as well as to develop new bioengineered tubes for the drainage of lymphedematous extremities.

1. Vaillant L, Tauveron V. [Primary lymphedema of limbs]. Presse Med. 2010;39(12):1279-86.
2. Lee JW, Lee TY, Moon KC, You HJ, Kim DW. Lymphatic complex transfer as combined lymph vessel and node transfer for advanced stage upper extremity lymphedema. J Vasc Surg Venous Lymphat Disord. 2023.
3. Olszewski WL, Zaleska M. A novel method of edema fluid drainage in obstructive lymphedema of limbs by implantation of hydrophobic silicone tubes. J Vasc Surg Venous Lymphat Disord. 2015;3(4):401-8.
4. Kwon HR, Hwang JH, Mun GH, Hyun SH, Moon SH, Lee KH, et al. Predictive role of lymphoscintigraphy undergoing lymphovenous anastomosis in patients with lower extremity lymphedema: a preliminary study. BMC Med Imaging. 2021;21(1):188.
5. Nuri T, Iwanaga H, Otsuki Y, Ueda K. Lymphoscintigraphy for prediction of effect of lymphaticovenular anastomosis for treatment of secondary lower limb lymphedema. J Vasc Surg Venous Lymphat Disord. 2022;10(5):1079-86 e2.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb lymphedema (Grade II-IV)
* Total occlusion at lymphoscintigraphy
* Patients treated at Centro Hospitalar Universitário de São João by the same surgical team
* Age >18 years old;
* Lymphedema praecox
* Lower limb perimeter >15% superior to contralateral limb

Exclusion Criteria:

* Secondary lymphedema
* Congenital lymphedema (Milroy, Meige, Klinefelter, Noonan, and Turner syndromes)
* Acute infection of the limb
* Chronic venous insufficiency
* Neoplasic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower limb circumference in cm | Preoperative, six months, one year, second year
  Lower limb circumference in cm - ankle, calf 15 cm below the knee; knee; thigh 15 cm above the knee

SECONDARY OUTCOMES:
PROMS - Lymphedema quality of life | preoperative, six months, one year, two years
  diseae specific qol questionnaire
PROMS - SF 36 | preoperative, six months, one year, two years
  Qol questionnaire
Lymphoscintigraphy | preoperative, one year (only in the intervention group)
  diagnostic exam

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
only principal Investigators

REFERENCES:
- [Background] Olszewski WL, Zaleska M. A novel method of edema fluid drainage in obstructive lymphedema of limbs by implantation of hydrophobic silicone tubes. J Vasc Surg Venous Lymphat Disord. 2015 Oct;3(4):401-408. doi: 10.1016/j.jvsv.2015.05.001. Epub 2015 Jun 30. PMID 26992618
- [Background] Kwon HR, Hwang JH, Mun GH, Hyun SH, Moon SH, Lee KH, Choi JY. Predictive role of lymphoscintigraphy undergoing lymphovenous anastomosis in patients with lower extremity lymphedema: a preliminary study. BMC Med Imaging. 2021 Dec 8;21(1):188. doi: 10.1186/s12880-021-00713-1. PMID 34879819